CLINICAL TRIAL: NCT04240067
Title: Multimarker Approach for Acute Dyspnea in Elderly Patients Admitted in the Emergency Department
Acronym: READ-MA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/466
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2020-01

CONDITIONS: Acute Dyspnea; Acute Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Acute Heart Failure
  Interventions: Diagnostic Test: READ-MA Multimarker Approach
- No Acute Heart Failure
  Interventions: Diagnostic Test: READ-MA Multimarker Approach

INTERVENTIONS:
Diagnostic Test: READ-MA Multimarker Approach — The presence or absence of ALSHF (gold standard used in the READ study) : diagnosis by 2 experts (cardiologist and emergency physician) based on data collected in the ED and during hospitalization (clinical examination, history, usual treatment, haemodynamic parameters, ECG, chest X-ray, emergency treatment, clinical and paraclinical results during hospitalization), biological assays (except NT-proBNP) and echocardiography (Left Ventricular Ejection Fraction, segmental kinetic, potential valvulopathy, transmitral flow, tissue doppler E' velocity) performed by a cardiologist within 24 hours of admission.

SUMMARY:
Elderly people constitute the largest proportion of emergency department (ED) patients, representing 12% of all ED admissions. The need for diagnostic tests or therapeutic interventions is much greater in this patient population. Cardiovascular diseases and symptoms represent 12% of the causes for ED admission, and patients suffering from cardiovascular disease are those whose ED visit lasts longest.

The diagnostic approach in the ED in elderly patients admitted for acute dypsnoea is complex, and early identification of acute left-sided heart failure (ALSHF) is vital as it has an impact on prognosis. The clinical signs are difficult to interpret, and are non-specific, particularly at the acute phase and in elderly or obese patients. Indeed, some authors have reported up to 50% of diagnostic errors in elderly patients.

Measure of the blood concentration of a natriuretic peptide allows a quick diagnosis. However, peptides alone suffer from several limitations, particularly in situations that are often encountered in elderly patients, such as sepsis, renal failure, acute coronary syndrome, pulmonary embolism, chronic respiratory failure, atrial fibrillation and high body mass index. Diagnostic performance deteriorates with increasing age, and there is a significant increase in this grey-zone in patients aged ≥75 years. In critical situations in elderly patients, assessment of natriuretic peptides serve mainly to rule out a diagnosis of left heart failure.

Some authors have studied other biomarkers showing their performance in the diagnosis of ALSHF. These are biomarkers involved in remodeling and myocardial fibrosis (ST2, Galectin-3) or involved in myocardial injury (High-sensitivity Troponin-I).

Therefore, a combined "multimarker" approach could improve the diagnostic performance of ALSHF.

READ (NCT02531542) is a diagnostic study including patients over the age of 75 admitted to acute dyspnea in the ED, to demonstrate the superiority of an ultrasound protocol (the READ protocol) on NT-proBNP in the ALSHF diagnosis.

The hypothesis is that the diagnostic accuracy of a multimarker diagnostic approach, namely the READ-MA method, combining NT-proBNP, High-sensitivity Troponin-I, ST2 and Galectin-3 would be superior to that of NT-proBNP assessment for the diagnosis of ALSHF in elderly patients (≥75 years) admitted to the ED.

ELIGIBILITY:
Inclusion Criteria :

* Admission to the Emergency Department with age ≥ 75 years
* AND criteria of acute dyspnea :

Breathe rate ≥ 25 cycles/minute or PaO2 ≤ 70 mmHg or SpO2 ≤ 92% in room air or PacO2 ≥ 45 mmHg and pH ≤ 7.35

- AND Electrocardiogram in sinus rhythm or in atrial fibrillation at admission

Exclusion Criteria:

* none

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged ≥75 years admitted to the ED for acute dyspnea
Sampling Method: Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
To assess the diagnostic performance of the multimarker approach (combining NT-proBNP, High-sensitivity Troponin-I, ST2 and Galectin-3) for the diagnosis of ALSHF in patients aged ≥75 years admitted to the ED for acute dyspnea | 1 day
  1. The presence or absence of ALSHF (gold standard used in the READ study) : diagnosis by 2 experts (cardiologist and emergency physician) based on data collected in the ED and during hospitalization, biological assays (except NT-proBNP) and echocardiography performed by a cardiologist.
  2. The positivity of the evaluated test (multi-marker approach) :
     * For NT-proBNP, the threshold for positivity is higher than 1800 pg/mL. There is no consensus for High-Sensitivity Troponin-I, ST2 and Galectin-3. Firstly, the optimal threshold of each of these 3 biomarkers will be assessed by ROC curve, then the best combination between these 4 biomarkers will be tested to obtain an optimal discrimination (sensitivity, specificity positive and negative predictive values), positive and negative likelihood ratios) using various methods.

SECONDARY OUTCOMES:
To demonstrate the superiority of the multimarker approach (NT-proBNP, High-sensitivity Troponin-I, ST2 and Galectin-3) over NT-proBNP alone for the diagnosis of ALSHF in patients aged ≥75 years admitted to the ED for acute dyspnea | 1 day
  To demonstrate the superiority of this combined multi-marker approach combining NT-proBNP, Troponin-I ultrasensitive, ST-2 and Galectin-3 on NT-proBNP alone in the diagnosis of ALSHF in subjects over 75 years admitted to emergencies for acute dyspnea, will be evaluated :
  * The presence or absence of acute left heart failure (gold standard selected in the context of the READ study) will be determined using the previously defined criteria
  * The evaluated test will be the best multimarker approach previously determined, classified as positive or negative using the previously defined criteria
  * The comparative test (NT-proBNP alone) will be classified positive for a threshold higher than 1800 pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric MAUNY, Prof, MD, PhD, Study Chair — Centre Hospitalier Universitaire de Besancon; Noémie NMINEJ, Study Chair — Centre Hospitalier Universitaire de Besancon; Patrick RAY, Prof, MD, PhD, Study Chair — Centre Hospitalier Universitaire Dijon; Camille CHENEVIER-GOBEAUX, PharmD, PhD, Study Chair — Hôpital Cochin, Assistance Publique Hôpitaux de Paris; Marie-Hélène TOURNOYS, PharmD, Study Chair — Centre Hospitalier de Bethune; Marc PUYRAVEAU, MSc, Study Chair — Centre Hospitalier Universitaire de Besancon; Alain-Eric DUBART, MD, Study Chair — CH Béthune
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, Franche-Comté, France

IPD SHARING:
Plan to Share IPD: Undecided